CLINICAL TRIAL: NCT06982508
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Trial to Assess the Effects of Obicetrapib on Levels of Antioxidants in Plasma and HDL Particles in Healthy Volunteers: The VERMEER Study
Brief Title: Evaluation of Obicetrapib on Antioxidant Levels in Plasma and HDL Particles of Healthy Volunteers
Acronym: VERMEER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: MB Clinical Research and Consulting LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TA-8995-207
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Antioxidant Absorption
Keywords: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obicetrapib 10mg (Experimental)
  Interventions: Drug: Obicetrapib 10mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obicetrapib 10mg — Active Drug
  Arms: Obicetrapib 10mg
Drug: Placebo — Placebo Control
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Obicetrapib works to change antioxidant levels in HDL and plasma, as well as retinal tissue. The main questions it aims to answer are:

Do Obicetrapib effect absorption of antioxidants in a person's blood or their eye tissue? Researchers will compare Obicetrapib to a placebo (a look-alike substance that contains no drug) to see if Obicetrapib helps improve a person's ability to absorb antioxidants.

Participants will:

Take Obicetrapib or a placebo every day for 4 months Visit the clinic once every 8 weeks for checkups and tests Have their blood taken and their eyes checked to measure antioxidant levels

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity > 20/60 in both eyes with or without corrective lenses

Exclusion Criteria:

* Type 2 diabetes
* Active liver disease
* Any clinically significant macular pathology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sum of Percent Change of Antioxidant Levels within HDL | 16 Weeks
  The primary efficacy endpoint is the effect of obicetrapib on the sum of the percent changes in lutein, zeaxanthin, and α-tocopherol levels within HDL particles from baseline to visit 4 (week 16) compared to placebo.

SECONDARY OUTCOMES:
Effects of Obicetrapib on Percent Changes of Antioxidant Levels in Retinal Tissue, Plasma, and HDL Particles | 8 and 16 weeks
  The secondary efficacy endpoints are the effect of obicetrapib compared to placebo on the percent changes from baseline to visit 3 (week 8) and baseline to visit 4 (week 16) for the following variables:
  * MPOD
  * Plasma level of α-tocopherol
  * Plasma level of lutein
  * Plasma level of zeaxanthin
  * Lutein within HDL particles
  * Zeaxanthin within HDL particles
  * α-tocopherol within HDL particles
  * Sum of the percent changes in lutein, zeaxanthin, and α-tocopherol in plasma
  * Sum of the percent changes in lutein, zeaxanthin, and α-tocopherol within HDL particles from baseline to visit 3 (week 8)
  * LDL-C
  * HDL-C
  * Non-HDL-C
  * ApoA1
  * ApoB
  * Lp(a)
  * TC
  * TG

CONTACTS AND LOCATIONS:
Locations (1):
- Excellence Medical Research, Miami Gardens, Florida, United States